CLINICAL TRIAL: NCT06037564
Title: Booster-free Antiretroviral Therapy for Persons Living With HIV and Multidrug Resistance: A Multicentre Multi-stage Randomized Trial
Brief Title: B-free Multistage Trial
Acronym: B-free
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-free trial - Stage 1
Record Dates: First submitted 2023-04-24; First posted 2023-09-14 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: HIV; Drug Resistance; Drug Drug Interaction
Keywords: HIV; Doravirine; Dolutegravir; Drug resistance; Drug-drug interaction
MeSH Terms: interventions — doravirine; dolutegravir; Lamivudine

STUDY DESIGN:
Intervention Model Description: Multi-stage, randomized, multicenter, open-label non-inferiority trial with active control
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Doravirine 100 mg (Pifeltro®) will be administered once daily in combination with co-formulated dolutegravir/lamivudine 50/300 mg (Dovato®) for a duration of 48 weeks.
  Interventions: Drug: DOR/DTG/3TC
- Control (No Intervention): Participants randomized to the control arm will continue to take their fully suppressive ART at baseline. The following selection of treatment combinations could be encountered in the control group (among others):
  * Once-daily co-formulated elvitegravir 150 mg, cobicistat 150 mg, tenofovir alafenamide 10 mg, emtricitabine 200 mg (Genvoya®) and darunavir 800 mg (e.g. Darunavir Mylan®)
  * Once-daily co-formulated darunavir 800 mg, cobicistat 150 mg, tenofovir alafenamide 10 mg, emtricitabine 200 mg (Symtuza ®) and DTG 50 mg (Tivicay ®)
  * Once-daily DTG 50 mg (Tivicay®), darunavir 800 mg (e.g. Darunavir Mylan®), and ritonavir 100 mg (Norvir®)
  * Etravirine 200 mg twice daily (Intelence®), raltegravir 400 mg twice daily (Isentress®),darunavir 800 mg once daily (e.g. Darunvair Mylan®) and ritonavir 100 mg once daily (Norvir®)

INTERVENTIONS:
Drug: DOR/DTG/3TC — Doravirine 100 mg (Pifeltro®) will be administered once daily in combination with co-formulated dolutegravir/lamivudine 50/300 mg (Dovato®) for a duration of 48 weeks.
  Other Names: Doravirine (Pifeltro®) + Dolutegravir/Lamivudine (Dovato®)
  Arms: Intervention

SUMMARY:
The primary objective of the study is to evaluate the efficacy of a booster-free regimen including DOR/DTG/3TC among HIV-suppressed PLWH with previous virological failure. The key secondary objectives are i) to determine whether switching to DOR / DTG / 3TC leads to lower burden of DDI compared to continuing a booster-containing regimen, and ii) to assess changes in patient perception on treatment acceptability and satisfaction, as well as health-related quality of life after a switch to booster-free ART.

Qualitative sub-study:

Qualitative objectives will be met using semi-structured interviews. Thirty people (15 from the intervention arm, 15 from the control arm) will be interviewed twice, at week 0 and week 48. Additional 15 individuals from the observational cohort will be interviewed once. Interviews will take place following study visits and performed using semi-structured guides. The guide for the interviews at week 48 will be based on results from analyses of the interviews conducted at week 0.

DETAILED DESCRIPTION:
Life expectancy of persons living with HIV on antiretroviral therapy (ART) is increasing and drug-drug interactions (DDI) with co-medications are becoming a major concern. Individuals who previously experienced virological failure are at risk of DDI as they are generally treated with ritonavir- or cobicistat-boosted ART. The high potency as well as the favorable safety and pharmacokinetic profile of new antiretroviral drugs, including dolutegravir (DTG) and doravirine (DOR), support their evaluation as part of un-boosted therapy for individuals with a history of virological failure. In this adaptive trial within the Swiss HIV Cohort Study (SHCS) and partner clinics in the Netherlands, the investigators aim to evaluate the efficacy and acceptability of the booster-free regimen DOR/DTG/3TC for treatment-experienced individuals.

ELIGIBILITY:
Inclusion criteria

* Informed consent as documented by signature
* Age ≥18 years
* Documented HIV-1 infection
* On ART including a pharmacological booster (ritonavir or cobicistat) and at least 2 drugs from classes other than NRTI (e.g. non-nucleoside reverse transcriptase inhibitor, integrase-inhibitor, protease inhibitor or entry inhibitor)
* History of ART change due to virological failure
* HIV-RNA <50 cp/mL at screening and for at least 24 weeks before screening, one blip with less than 200 cp/mL allowed

Exclusion criteria

* Creatinine clearance <30mL/min, calculated using the CKD-EPI formula
* Known hypersensitivity, allergy, or intolerance to DOR, DTG, or 3TC
* Presence of major drug resistance mutations against DTG (G118R, G140R, Q148H, Q148K, Q148R, R263K) or DOR (V106A, Y188L, F227C, F227L, M230L, Y318F) according to IAS-USA in individual cumulative resistance analyses. Patients without available resistance testing should not be excluded if no resistance to DTG and/or DOR is assumed based on ART history.
* Concomitant use of drugs that decrease DTG or DOR blood concentrations
* Chronic hepatitis B infection, defined as a positive hepatitis B surface antigen (HBsAg) at the screening visit
* Women who are pregnant or breast-feeding. Women of childbearing potential (women who are not surgically sterilized / hysterectomised and / or post-menopausal for longer than 2 years must have a negative pregnancy test at screening).
* Participation in another ART intervention study within the 30 days preceding and during the present study.

Qualitative sub-study

The same inclusion and exclusion criteria as those listed above will be applied. Fifteen persons who were excluded from the trial based on the exclusion criteria above will be recruited for qualitative interviews. In addition to the criteria mentioned above, individuals who are not fluent in German or French will be excluded from the qualitative sub-study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Loss of viral suppression | Week 48
  Difference in the proportion of individuals with an HIV-RNA ≥50 cp/mL at 48 weeks between the treatment arms.

SECONDARY OUTCOMES:
Changes in DDI score from week 0 to 48 | Week 0 and 48
  Using the University of Liverpool Drug Database (https://www.hiv-druginteractions.org/), the prescribed ART and co-medications will be categorized as red flag (3 points) for severe DDIs when co-administration is contraindicated, amber flag (2 points) for potential clinically significant DDIs manageable by dose adjustment or clinical monitoring, yellow flag (1 point) for DDIs of weak clinical relevance with no need of a priori dosage adjustment or monitoring, and a green flag (0 points) for no interactions. Amber flag DDIs will be downgraded to 1 point if there is evidence that the DDI was managed correctly (i.e. DTG administered 2 hours before or 6 hours after taking divalent cations). The sum of all points at visit 6, week 48 will be compared to baseline.
Patient report outcomes concerning changes in treatment satisfaction between baseline and 48 weeks, as determined using the HIV Treatment Satisfaction Questionnaire HIVTSQc (change version). | Week 0 to 48
  The investigators will assess changes in treatment satisfaction between week 0 and 48 using the validated HIV Treatment Satisfaction Questionnaire HIVTSQc (change version).
Proportion of patients experiencing confirmed virological failure | Week 48
  Proportion of patients experiencing confirmed virological failure, defined as 2 consecutive plasma HIV viral loads ≥200 copies/mL
Proportion of individuals detected with new drug resistance | Week 0 to 48
  Proportion of individuals experiencing impairment / loss of future drug options throughout the study period, defined as new detection of resistance-associated mutations against DOR, DTG, 3TC (intervention-arm) or against the components of the ART regimen that the virus was considered to be sensitive to at randomization (based on historic resistance testing or treatment history; control-arm).
Proportion of individuals with any moderate (orange flag) or severe (red flag) DDI | Week 0 to 48
  Proportion of individuals with any moderate (orange flag) or severe (red flag) DDI at any study visit between baseline and week 48, based on the results from the Liverpool drug interaction database (www.hiv-druginteractions.org).
Proportion of patients with DDI leading to suboptimal management of comorbidities | Week 0 and 48
  Proportion of patients with DDI leading to suboptimal management of comorbidities between baseline and week 48, as reported by the cohort physician.
Patient report outcomes concerning differences in quality of life between both groups at week 48 assessed by the World Health Organization Quality-of-Life- HIV Bref (WHOQOL-HIV BREF) questionnaire | Week 48
  Differences in quality of life between both groups at week 48, assessed using the World Health Organization Quality-of-Life- HIV Bref (WHOQOL-HIV BREF) questionnaire
Patient report outcomes concerning differences in treatment satisfaction between both groups assessed by HIV Treatment Satisfaction Questionnaires | Week 48
  The investigators will assess the differences in treatment satisfaction between both groups at week 48, as determined using the validated HIV Treatment Satisfaction Questionnaires HIVTSQ.
Proportion of individuals reporting depression assessed by Patient Health Questionnaire-9 | Week 0 and 48
  Depression will be assessed at baseline and week 48, assessed using the Patient Health Questionnaire-9 (PHQ-9)
Changes in intact proviral HIV-DNA levels | Week 0 to 48
  Changes in intact proviral HIV-DNA levels in peripheral blood mononuclear cells (PBMCs) between baseline and week 48. Stored PBMC samples will be used to determine HIV-DNA levels by a digital droplet PCR (ddPCR) assay using the RAINDANCE system.
Proportion of individuals who develop a detectable HBV viral load | Weeks 24 and 48
  Proportion of individuals with a positive anti-HBc and negative anti-HBs ("anti-HBc alone") who develop a detectable HBV viral load (>50 IU/mL) at weeks 24 and 48.
Cumulative cost of all ART drugs used | Week 0 to 48
  The 48-weeks cumulative cost of the received ART regimen will be calculated using prices published by the Federal Office of Public Health (https://www.spezialitaetenliste.ch/ShowPreparations.aspx).
Perception of the trial and/or of HIV-related research in general assessed by qualitative interviews in a subset of approximately 30 trial participants | Week 0 and 48
  Perception of the trial and/or of HIV-related research in general.
Acceptability conditions of participation in the trial assessed by qualitative interviews in a subset of approximately 30 trial participants | Week 0 and 48
  Acceptability conditions, understood as all barriers and facilitators to be involved in a trial.
Needs regarding the booster-free regimen or regarding ART in general assessed by qualitative interviews in a subset of approximately 30 trial participants | Week 0 and 48
  Needs regarding the booster-free regimen or regarding ART in general for participants included in the observational cohort.
Expectations regarding the booster-free regimen or regarding ART in general assessed by qualitative interviews in a subset of approximately 30 trial participants | Week 0 and 48
  Expectations regarding the booster-free regimen or regarding ART in general for participants included in the observational cohort.
Perspectives on how the participants' current and anticipated needs can be assessed by qualitative interviews in a subset of approximately 30 trial participants | Week 0 and 48
  Perspectives on how the participants' current and anticipated needs can be addressed by research.

OTHER OUTCOMES:
Change in CD4 cell count from baseline to week 48 | Week 0 and 48
  The CD4 cell counts will be obtained at baseline and week 48.
Change in metabolic variables (cholesterol) | Week 0 and 48
  Change in total cholesterol
Change in metabolic variables (low density lipoprotein) | Week 0 and 48
  Change in low density lipoprotein-cholesterol
Change in metabolic variables (high density lipoprotein) | Week 0 and 48
  Change in high density lipoprotein-cholesterol
Change in metabolic variables (triglycerides) | Week 0 and 48
  Change in triglycerides
Change in body weight | Week 0 and 48
  Change in body weight from baseline to week 48
Change in BMI | Week 0 and 48
  Change in BMI from baseline to week 48
Change in renal function, assessed by glomerular filtration rate | Week 0 and 48
  Changes in glomerular filtration rate (calculated using the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] formula) from baseline to week 48
Change in renal function, assessed by urine protein-to-creatinine ratio | Week 0 and 48
  Change in renal function (glomerular filtration rate) using the urine protein-to-creatinine ratio from baseline to week 48
Proportion of patients with new drug-related CNS symptom(s) at week 4 | Week 4
  Proportion of patients with new drug-related central nervous system (CNS) symptom(s) at the 4 week visit.
Proportion of patients with new drug-related CNS symptom(s) reporting new drug-related CNS symptom(s) at any time point between baseline and week 48. | Week 0 to 48
  Occurrence of CNS Adverse Events (AEs) in patients new to DTG
Proportion of patients with a Serious Adverse Event (SAE) at any time point | Week 0 to 48
  Proportion of patients with a SAE, graded using the Division of AIDS table for grading AEs at any time point.

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Wandeler, Prof, Principal Investigator — Inselspital, Bern, Switzerland
Locations (8):
- Switzerland (8):
  - Cantonal Hospital Aarau, Aarau, Canton of Aargau
  - University Hospital Basel, Basel
  - Inselgruppe AG, Bern
  - University Hospital Geneva, Geneva
  - University of Lausanne Hospitals, Lausanne
  - Lugano Regional Hospital Lugano, Lugano
  - Cantonal Hospital of St. Gallen, Sankt Gallen
  - University Hospital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ballif M, Braun D, Calmy A, Bernasconi E, Cavassini M, Tissot F, Stoeckle M, Schmid P, Fux CA, Van der Valk M, Brinkman K, Mudrikova T, Bonnet F, Leleux O, Saude M, Hirter D, Schwab N, Limacher A, Rintelen F, Kouyos R, Haerry D, Zambrano SC, Egloff M, Akre C, Peytremann-Bridevaux I, Rauch A, Wandeler G, Surial B. Booster-free anti-retroviral therapy for persons living with HIV and multidrug resistance (B-Free): protocol for a multicentre, multistage, randomised, controlled, non-inferiority trial. BMJ Open. 2024 Nov 21;14(11):e094912. doi: 10.1136/bmjopen-2024-094912. PMID 39578038